CLINICAL TRIAL: NCT00006304
Title: Pediatric Late Outcomes Protocol
Brief Title: Long-Term Effects of HIV Exposure and Infection in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG 219C; ACTG 219; PACTG 219C; 11196 (Registry Identifier: DAIDS ES); NCT00000786 (obsolete NCT alias)
Record Dates: First submitted 2000-09-27; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

SUMMARY:
As new drugs and vaccines are developed to prevent HIV disease progression and prolong survival of HIV infected patients, the short-term safety and effectiveness of these treatments are evaluated in research studies. However, the long-term effects, whether they are benefits or side effects, need to be studied as well. These long-term effects may have a greater impact on infants and children who are still growing and developing. The purpose of this study is to follow HIV-exposed and HIV infected infants, children, and adolescents who are seen at Pediatric AIDS Clinical Trials Group (PACTG) study sites. These patients will be observed for long-term benefits or any late harmful effects of medications or vaccines.

DETAILED DESCRIPTION:
The potential long-term benefits, toxicities, and other adverse outcomes of new anti-HIV therapies cannot be assessed within the time frame of most clinical trials. There is a need to better assess both positive and negative late outcomes and late treatment effects in growing children. This prospective, longitudinal study will evaluate the effects and their impact on children.

Children in this study will include patients who are HIV infected, were exposed to HIV or anti-HIV drugs prior to or at the time of their birth, or children of patients followed at Pediatric AIDS Clinical Trial Group (PACTG) sites. Children will have a study visit every 3 months through the first year of life. After age 1, children who are HIV infected will continue to have study visits every 3 months, while children who are HIV uninfected will have study visits once a year. Study assessments will include complete physical exam, medical history, Tanner staging, neurologic exam, growth and quality of life assessments, and laboratory tests such as hematology, chemistries, and urinalysis. Not all assessments will be performed at each study visit. Patients will be followed until age 24.

ELIGIBILITY:
Inclusion Criteria

* Age 21 or younger (consent of parent or guardian required if under 18).
* Meet 1 of the following 3 requirements: 1) enrolled in a previous version of this study; 2) perinatally exposed to HIV, HIV vaccines, or antiretroviral treatment (must enroll before first birthday); 3) HIV infected infants, children, and adolescents (and their offspring) followed at PACTG sites.

Exclusion Criteria

* Unable to adhere to study visit schedules.

Ages: 24 Hours to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4150
Dates: Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Oleske, Study Chair; Michael Brady, Study Chair; Wayne Dankner, Study Chair
Locations (92):
- United States (89):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - UCLA Med Ctr / Pediatrics, Los Angeles, California
  - UCLA Med Ctr, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Sacred Heart Children's Hosp / CMS of Florida, Pensacola, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Univ of South Florida, St. Petersburg, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Earl K Long Early Intervention Clinic, New Orleans, Louisiana
  - Univ Hosp, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Childrens Hospital of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - St. Louis Children's Hosp, St Louis, Missouri
  - Cooper Hosp, Camden, New Jersey
  - Robert Wood Johnson AIDS Program, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Montefiore Medical / AECOM, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Oregon Health Sciences Univ, Portland, Oregon
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Brady MT, Clark C, Weedy C, Fowler M, Mofenson L, Oleske J. Disclosure of HIV diagnosis to children in ACTG clinical trials (ACTG 219). Int Conf AIDS. 1996 Jul 7-12;11(2):43 (abstract no WeD131)
- [Background] Gaughan DM, Mofeson LM, Hughes MD, Seage GR, Oleske JM. Avascular necrosis of the hip (Leggs-Calve-Perthes disease [LCPD]) in HIV-infected children in long-term follow-up: PACTG study 219. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 638)
- [Background] Buchacz K, Cervia JS, Lindsey JC, Hughes MD, Seage GR 3rd, Dankner WM, Oleske JM, Moye J. Impact of protease inhibitor-containing combination antiretroviral therapies on height and weight growth in HIV-infected children. Pediatrics. 2001 Oct;108(4):E72. doi: 10.1542/peds.108.4.e72. PMID 11581480
- [Result] Culnane M, Fowler M, Lee SS, McSherry G, Brady M, O'Donnell K, Mofenson L, Gortmaker SL, Shapiro DE, Scott G, Jimenez E, Moore EC, Diaz C, Flynn PM, Cunningham B, Oleske J. Lack of long-term effects of in utero exposure to zidovudine among uninfected children born to HIV-infected women. Pediatric AIDS Clinical Trials Group Protocol 219/076 Teams. JAMA. 1999 Jan 13;281(2):151-7. doi: 10.1001/jama.281.2.151. PMID 9917118
- [Result] Gaughan DM, Mofenson LM, Hughes MD, Seage GR 3rd, Ciupak GL, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Osteonecrosis of the hip (Legg-Calve-Perthes disease) in human immunodeficiency virus-infected children. Pediatrics. 2002 May;109(5):E74-4. doi: 10.1542/peds.109.5.e74. PMID 11986480
- [Result] Hanson IC, Antonelli TA, Sperling RS, Oleske JM, Cooper E, Culnane M, Fowler MG, Kalish LA, Lee SS, McSherry G, Mofenson L, Shapiro DE. Lack of tumors in infants with perinatal HIV-1 exposure and fetal/neonatal exposure to zidovudine. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Apr 15;20(5):463-7. doi: 10.1097/00042560-199904150-00008. PMID 10225228
- [Result] Gaughan DM, Hughes MD, Seage GR 3rd, Selwyn PA, Carey VJ, Gortmaker SL, Oleske JM. The prevalence of pain in pediatric human immunodeficiency virus/acquired immunodeficiency syndrome as reported by participants in the Pediatric Late Outcomes Study (PACTG 219). Pediatrics. 2002 Jun;109(6):1144-52. doi: 10.1542/peds.109.6.1144. PMID 12042556
- [Result] Gortmaker SL, Hughes M, Cervia J, Brady M, Johnson GM, Seage GR 3rd, Song LY, Dankner WM, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Effect of combination therapy including protease inhibitors on mortality among children and adolescents infected with HIV-1. N Engl J Med. 2001 Nov 22;345(21):1522-8. doi: 10.1056/NEJMoa011157. PMID 11794218
- [Result] Howland LC, Gortmaker SL, Mofenson LM, Spino C, Gardner JD, Gorski H, Fowler MG, Oleske J. Effects of negative life events on immune suppression in children and youth infected with human immunodeficiency virus type 1. Pediatrics. 2000 Sep;106(3):540-6. doi: 10.1542/peds.106.3.540. PMID 10969100
- [Result] Nucleoside exposure in the children of HIV-infected women receiving antiretroviral drugs: absence of clear evidence for mitochondrial disease in children who died before 5 years of age in five United States cohorts. J Acquir Immune Defic Syndr. 2000 Nov 1;25(3):261-8. doi: 10.1097/00126334-200011010-00009. PMID 11115957
- [Result] Gaughan DM, Hughes MD, Oleske JM, Malee K, Gore CA, Nachman S; Pediatric AIDS Clinical Trials Group 219C Team. Psychiatric hospitalizations among children and youths with human immunodeficiency virus infection. Pediatrics. 2004 Jun;113(6):e544-51. doi: 10.1542/peds.113.6.e544. PMID 15173535
- [Result] Farley J, Gona P, Crain M, Cervia J, Oleske J, Seage G, Lindsey J; Pediatric AIDS Clinical Trials Group Study 219C Team. Prevalence of elevated cholesterol and associated risk factors among perinatally HIV-infected children (4-19 years old) in Pediatric AIDS Clinical Trials Group 219C. J Acquir Immune Defic Syndr. 2005 Apr 1;38(4):480-7. doi: 10.1097/01.qai.0000139397.30612.96. PMID 15764965
- [Result] Kest H, Brogly S, McSherry G, Dashefsky B, Oleske J, Seage GR 3rd. Malignancy in perinatally human immunodeficiency virus-infected children in the United States. Pediatr Infect Dis J. 2005 Mar;24(3):237-42. doi: 10.1097/01.inf.0000154324.59426.8d. PMID 15750460
- [Result] Brogly S, Williams P, Seage GR 3rd, Oleske JM, Van Dyke R, McIntosh K; PACTG 219C Team. Antiretroviral treatment in pediatric HIV infection in the United States: from clinical trials to clinical practice. JAMA. 2005 May 11;293(18):2213-20. doi: 10.1001/jama.293.18.2213. PMID 15886376
- [Result] Gona P, Van Dyke RB, Williams PL, Dankner WM, Chernoff MC, Nachman SA, Seage GR 3rd. Incidence of opportunistic and other infections in HIV-infected children in the HAART era. JAMA. 2006 Jul 19;296(3):292-300. doi: 10.1001/jama.296.3.292. PMID 16849662
- [Result] Williams PL, Storm D, Montepiedra G, Nichols S, Kammerer B, Sirois PA, Farley J, Malee K; PACTG 219C Team. Predictors of adherence to antiretroviral medications in children and adolescents with HIV infection. Pediatrics. 2006 Dec;118(6):e1745-57. doi: 10.1542/peds.2006-0493. Epub 2006 Nov 13. PMID 17101712
- [Result] Sirois PA, Montepiedra G, Kapetanovic S, Williams PL, Pearson DA, Malee K, Garvie PA, Kammerer BL, Nichols SL, Nozyce ML, Mintz M, Mitchell WG, Oleske JM; IMPAACT/PACTG 219C Team. Impact of medications prescribed for treatment of attention-deficit hyperactivity disorder on physical growth in children and adolescents with HIV. J Dev Behav Pediatr. 2009 Oct;30(5):403-12. doi: 10.1097/dbp.0b013e3181ba0cf6. PMID 19827220
- [Result] Levin MJ, Anderson JP, Seage GR 3rd, Williams PL; PACTG/IMPAACT 219C Team. Short-term and long-term effects of highly active antiretroviral therapy on the incidence of herpes zoster in HIV-infected children. J Acquir Immune Defic Syndr. 2009 Feb 1;50(2):182-91. doi: 10.1097/QAI.0b013e31819550a4. PMID 19131890
- [Result] Edathodu J, Halim MM, Dahham MB, Alrajhi AA. Mother-to-child transmission of HIV: experience at a referral hospital in Saudi Arabia. Ann Saudi Med. 2010 Jan-Feb;30(1):15-7. doi: 10.4103/0256-4947.59367. PMID 20103953
- [Result] Kapetanovic S, Aaron L, Montepiedra G, Sirois PA, Oleske JM, Malee K, Pearson DA, Nichols SL, Garvie PA, Farley J, Nozyce ML, Mintz M, Williams PL; Pediatric AIDS Clinical Trials. The use of second-generation antipsychotics and the changes in physical growth in children and adolescents with perinatally acquired HIV. AIDS Patient Care STDS. 2009 Nov;23(11):939-47. doi: 10.1089/apc.2009.0121. PMID 19827949
- [Result] Nachman SA, Chernoff M, Gona P, Van Dyke RB, Dankner WM, Seage GR 3rd, Oleske J, Williams PL; PACTG 219C Team. Incidence of noninfectious conditions in perinatally HIV-infected children and adolescents in the HAART era. Arch Pediatr Adolesc Med. 2009 Feb;163(2):164-71. doi: 10.1001/archpedi.163.2.164. PMID 19188649
- [Result] Williams PL, Van Dyke R, Eagle M, Smith D, Vincent C, Ciupak G, Oleske J, Seage GR 3rd; PACTG 219C Team. Association of site-specific and participant-specific factors with retention of children in a long-term pediatric HIV cohort study. Am J Epidemiol. 2008 Jun 1;167(11):1375-86. doi: 10.1093/aje/kwn072. Epub 2008 Apr 15. PMID 18413359
- [Result] Lyon ME, Williams PL, Woods ER, Hutton N, Butler AM, Sibinga E, Brady MT, Oleske JM. Do-not-resuscitate orders and/or hospice care, psychological health, and quality of life among children/adolescents with acquired immune deficiency syndrome. J Palliat Med. 2008 Apr;11(3):459-69. doi: 10.1089/jpm.2007.0148. PMID 18363489
- [Result] Lindsey JC, Malee KM, Brouwers P, Hughes MD; PACTG 219C Study Team. Neurodevelopmental functioning in HIV-infected infants and young children before and after the introduction of protease inhibitor-based highly active antiretroviral therapy. Pediatrics. 2007 Mar;119(3):e681-93. doi: 10.1542/peds.2006-1145. Epub 2007 Feb 12. PMID 17296781
- [Result] Seage GR 3rd, Buchacz K, Weinberg GA, Patel K, McIntosh K, Dankner WM. The Pediatric AIDS Severity Score (PASS): a multidimensional AIDS-severity adjustment for pediatric HIV infection. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):603-10. doi: 10.1097/01.qai.0000242453.20521.4f. PMID 17003692
- [Result] Williams PL, Marino M, Malee K, Brogly S, Hughes MD, Mofenson LM; PACTG 219C Team. Neurodevelopment and in utero antiretroviral exposure of HIV-exposed uninfected infants. Pediatrics. 2010 Feb;125(2):e250-60. doi: 10.1542/peds.2009-1112. Epub 2010 Jan 18. PMID 20083530
- [Result] Malee K, Williams PL, Montepiedra G, Nichols S, Sirois PA, Storm D, Farley J, Kammerer B; PACTG 219C Team. The role of cognitive functioning in medication adherence of children and adolescents with HIV infection. J Pediatr Psychol. 2009 Mar;34(2):164-75. doi: 10.1093/jpepsy/jsn068. Epub 2008 Jul 22. PMID 18647794
- [Result] Kapetanovic S, Aaron L, Williams PL, Farley J, Sirois PA, Garvie PA, Pearson DA, Oleske JM, Montepiedra G; The IMPAACT PACTG 219C Team. Relationships between the use of second-generation antipsychotics and changes in total cholesterol levels in children and adolescents perinatally infected with HIV. Neurobehav HIV Med. 2010 Aug;2010(2):39-48. doi: 10.2147/NBHIV.S12517. PMID 20865061
- [Result] Malee K, Williams P, Montepiedra G, McCabe M, Nichols S, Sirois PA, Storm D, Farley J, Kammerer B; PACTG 219C Team. Medication adherence in children and adolescents with HIV infection: associations with behavioral impairment. AIDS Patient Care STDS. 2011 Mar;25(3):191-200. doi: 10.1089/apc.2010.0181. Epub 2011 Feb 16. PMID 21323533